CLINICAL TRIAL: NCT03500471
Title: Safety and Feasibility Between Robotic and Laparoscopic Total Gastrectomy With D2 Lymphadenectomy for Locally Advanced Gastric Cancer：A Prospective Cohort Study
Brief Title: Robotic and Laparoscopic Total Gastrectomy With D2 Lymphadenectomy for Locally Advanced Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Yan Shi, Deputy director, Southwest Hospital, China
Other Study IDs: 20180108
Record Dates: First submitted 2018-03-28; First posted 2018-04-18 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer
Keywords: Laparoscopic; Robotic; Total Gastrectomy; AGC
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Experimental: Robotic surgery: Robotic-assisted Total Gastrectomy with D2 Lymphadenectomy
  Interventions: Procedure: Robotic-assisted Total Gastrectomy
- Compared: Laparoscopic surgery: Laparoscopic-assisted Total Gastrectomy with D2 Lymphadenectomy
  Interventions: Procedure: Laparoscopic-assisted Total Gastrectomy

INTERVENTIONS:
Procedure: Robotic-assisted Total Gastrectomy — Robotic-assisted total gastrectomy with D2 lymph node dissection will be performed with curative treated intent according to the patients' or their legal representatives'willing to choose robotic-assisted total gastrectomy and exclusing T4b、bulky lymph nodes or distant metastasis case by diagnostic laparoscopy. The alimentary canal reconstruction method is selected as esophageal jejunal R-Y anastomosis. Whether to reinforce the anastomotic manually is decided by the surgeon's experience. The reconstruction can be carried out by extracorporeal or intracorporeal anastomosis.
  Groups: Experimental: Robotic surgery
Procedure: Laparoscopic-assisted Total Gastrectomy — Laparoscopic-assisted total gastrectomy with D2 lymph node dissection will be performed with curative treated intent according to the patients' or their legal representatives'willing to choose laparoscopic-assisted total gastrectomy and exclusing T4b、bulky lymph nodes or distant metastasis case by diagnostic laparoscopy. The alimentary canal reconstruction method is selected as esophageal jejunal R-Y anastomosis. Whether to reinforce the anastomotic manually is decided by the surgeon's experience. The reconstruction can be carried out by extracorporeal or intracorporeal anastomosis.
  Groups: Compared: Laparoscopic surgery

SUMMARY:
This study is a prospective, single-center, non-randomized, controlled, non-blind, and non-inferiority observation trial comparing robotic-assisted total gastrectomy with D2 lymph nodal dissection for locally advanced gastric cancer patients with laparoscopic procedure.

DETAILED DESCRIPTION:
Since Kitano firstly reported laparoscopy-assisted distal gastrectomy in 1994, the number of patients undergoing the laparoscopic procedure has gradually increased. The latest Japanese gastric cancer treatment guideline recommends laparoscopic gastrectomy (LG) as an optional treatment for cStage Ⅰ gastric cancer (GC).

Based on the experience of early GC, most experienced surgeons have applied the laparoscopic procedure in patients with locally advanced gastric cancer (AGC) especially in east world like China, Japan and Korea. Though applying laparoscopic-assisted total gastrectomy (LATG) is much more difficulty than that of distal gastrectomy (DG), there are a mount of centers reported their experiences of this procedure. A meta-analysis including seventeen studies of 2313 patients (955 in LATG and 1358 in open total gastrectomy) demonstrated that LATG can have less blood loss, fewer analgesic uses, earlier passage of flatus, quicker resumption of oral intake, earlier hospital discharge, and reduced postoperative morbidity. However, the number of harvested lymph nodes, proximal resection margin, hospital mortality, 5-year OS and DFS were similar in both groups. According to the existing reports, LATG is technically safety and feasibility.

To overcome the limitations of laparoscopic surgery, robot systems have been introduced to treat GC providing technical advantages since Hashizume firstly reported. Yoon and Son respectively compared robot-assisted total gastrectomy (RATG) with LATG, they drew a common conclusion that the number of dissected lymph nodes and postoperative complications were similar in both groups. But Son found that the mean numbers of retrieved LNs along the splenic artery from RATG was higher than LATG (2.3 vs. 1.0, p = 0.013), as was also the case at the splenic hilum and artery (3.6 vs.1.9, p = 0.014). Regretfully, most of their reported cases were early gastric cancer (EGC). Other literatures reported AGC patients under RATG or LATG together with distal gastrectomy (DG), we haven't found any literature compare RATG with LATG alone for AGC retrospectively.

Since most literatures are EGC patients and retrospectively researches, we can't insist that patients with AGC may benefit under RATG. Therefore, we launch this prospective, single-center, non-randomized, controlled, non-blind, and non-inferiority observation trial comparing RATG for locally advanced gastric cancer patients with LATG.In the process of research,it will be divided into two groups according to the willing of patients or their legal representatives who choose one of the two procedures(RATG or LATG) to cure GC.The primary objective of this study is to assess whether RATG is comparable to laparoscopic approach in terms of overall postoperative morbidity rates. The secondary research objectives are to compare robotic with laparoscopic approach in terms of surgical outcomes, postoperative recovery courses.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven gastric adenocarcinoma;
2. Age: older than 18 years old, younger than 80 years old;
3. Tumor located in the upper third of the stomach or esophagogastric junction or other location, and is possible to be curatively resected by total gastrectomy;
4. Preoperative stage of cT2-4aN0-3M0 according to American Joint Committee on Cancer/Union for International Cancer Control 8th edition;
5. American Society of Anesthesiology (ASA) score of class I to III;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. Patients who freely give informed consent to participate in the clinical study;

Exclusion Criteria:

1. Early gastric cancer;
2. Age: younger than 18 years old, older than 80 years old;
3. Total gastrectomy with D2 lymphadenectomy was not required;
4. Enlarged or bulky regional lymph node diameter larger than 3 cm based on preoperative imaging;
5. Emergency surgery for gastric cancer-related complications (bleeding or complete obstruction or perforation);
6. Previous upper abdominal surgery (except laparoscopic cholecystectomy);
7. Previous neoadjuvant chemotherapy or radiotherapy for gastric cancer;
8. Unstable angina or myocardial infarction within the past 6 months;
9. Cerebrovascular accident within the past 6 months;
10. American Society of Anesthesiology (ASA) score of class more than III;
11. Severe respiratory disease (FEV1< 50%);
12. Continuous systemic steroid therapy within 1 month before the study;
13. Pregnant or breast-feeding women;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gastric cancer who need to received total gastrectomy with D2 lymphadenectomy.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Overall postoperative morbidity and mortality | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.

SECONDARY OUTCOMES:
Time of operation | 1 day
  The total time of operation
Estimated blood loss | 1 day
  Blood loss during intraoperative including the volume of negative pressure drainage bottle and the increasing weight of gauzes （ml）
Blood transfusion | 1 day
  Blood transfusion during operation
Length of proximal and distal cutting margin | 1 day
  Length of proximal and distal cutting margin of the specimen
Number of retrieved lymph nodes | 7 days
  Total number of harvested perigastric lymph node
Time to flatus | 30 days
  Time of anus exsufflation
Time to first ambulation | 30 days
  Time to walking about
Time to liquid diet | 30 days
  Time to liquid diet
Time to soft diet | 30 days
  Time to soft diet
Duration of postoperative hospital stay | 30 days
  Time from operation to hospital discharge
cost | 30days
  All costs of hospitalization

OTHER OUTCOMES:
3-year Overall survival rate | 3 years
  3-year Overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Peiwu Yu, M.D., Study Chair — Southwest Hospital, China
Locations (1):
- Department of General Surgery and Center of Microinvasive Gastrointestinal Surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Background] Haverkamp L, Weijs TJ, van der Sluis PC, van der Tweel I, Ruurda JP, van Hillegersberg R. Laparoscopic total gastrectomy versus open total gastrectomy for cancer: a systematic review and meta-analysis. Surg Endosc. 2013 May;27(5):1509-20. doi: 10.1007/s00464-012-2661-1. Epub 2012 Dec 14. PMID 23263644
- [Background] Etoh T, Honda M, Kumamaru H, Miyata H, Yoshida K, Kodera Y, Kakeji Y, Inomata M, Konno H, Seto Y, Kitano S, Hiki N. Morbidity and mortality from a propensity score-matched, prospective cohort study of laparoscopic versus open total gastrectomy for gastric cancer: data from a nationwide web-based database. Surg Endosc. 2018 Jun;32(6):2766-2773. doi: 10.1007/s00464-017-5976-0. Epub 2017 Dec 7. PMID 29218676
- [Background] Yoon HM, Kim YW, Lee JH, Ryu KW, Eom BW, Park JY, Choi IJ, Kim CG, Lee JY, Cho SJ, Rho JY. Robot-assisted total gastrectomy is comparable with laparoscopically assisted total gastrectomy for early gastric cancer. Surg Endosc. 2012 May;26(5):1377-81. doi: 10.1007/s00464-011-2043-0. Epub 2011 Nov 16. PMID 22083338
- [Background] Son T, Lee JH, Kim YM, Kim HI, Noh SH, Hyung WJ. Robotic spleen-preserving total gastrectomy for gastric cancer: comparison with conventional laparoscopic procedure. Surg Endosc. 2014 Sep;28(9):2606-15. doi: 10.1007/s00464-014-3511-0. Epub 2014 Apr 3. PMID 24695982
- [Background] Shen W, Xi H, Wei B, Cui J, Bian S, Zhang K, Wang N, Huang X, Chen L. Robotic versus laparoscopic gastrectomy for gastric cancer: comparison of short-term surgical outcomes. Surg Endosc. 2016 Feb;30(2):574-580. doi: 10.1007/s00464-015-4241-7. Epub 2015 Jul 25. PMID 26208497
- [Background] Pan HF, Wang G, Liu J, Liu XX, Zhao K, Tang XF, Jiang ZW. Robotic Versus Laparoscopic Gastrectomy for Locally Advanced Gastric Cancer. Surg Laparosc Endosc Percutan Tech. 2017 Dec;27(6):428-433. doi: 10.1097/SLE.0000000000000469. PMID 29211699
- [Background] Junfeng Z, Yan S, Bo T, Yingxue H, Dongzhu Z, Yongliang Z, Feng Q, Peiwu Y. Robotic gastrectomy versus laparoscopic gastrectomy for gastric cancer: comparison of surgical performance and short-term outcomes. Surg Endosc. 2014 Jun;28(6):1779-87. doi: 10.1007/s00464-013-3385-6. Epub 2014 Jan 3. PMID 24385251
- [Background] Wang W, Zhang X, Shen C, Zhi X, Wang B, Xu Z. Laparoscopic versus open total gastrectomy for gastric cancer: an updated meta-analysis. PLoS One. 2014 Feb 18;9(2):e88753. doi: 10.1371/journal.pone.0088753. eCollection 2014. PMID 24558421

DOCUMENTS (2):
  • Study Protocol (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03500471/Prot_000.pdf
  • Informed Consent Form (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03500471/ICF_001.pdf